CLINICAL TRIAL: NCT03721224
Title: Psychiatric Disorders and Clinical Features of Children With Psychogenic Cough
Brief Title: Psychiatric Disorders in Children With Psychogenic Cough
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Abdurrahman Cahid Örengül, Assistant Professor, Bezmialem Vakif University
Other Study IDs: BVU Psychogenic cough study 1
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Psychogenic Cough
Keywords: psychiatry, children, habit cough
MeSH Terms: conditions — somatic cough syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with psychogenic cough: children who were examined by Pediatric Respiratory Disease specialist and diagnosed as having a psychogenic cough.
  Interventions: Diagnostic Test: Kiddie Schedule for Affective Disorders and Schizophrenia
- control subjects: children who were referred to pediatrics clinics and do not have a chronical disease.
  Interventions: Diagnostic Test: Kiddie Schedule for Affective Disorders and Schizophrenia

INTERVENTIONS:
Diagnostic Test: Kiddie Schedule for Affective Disorders and Schizophrenia — Both of the clinical and control group will be evaluated via Psychiatric semi-structured interview

SUMMARY:
The study aims to evaluate psychiatric disorders and clinical features of children with psychogenic cough. Psychiatric disorders are assessed via a semi-structured interview (Kiddie Schedule for Affective Disorders and Schizophrenia) and clinical features are investigated via sociodemographic form, which was developped by researchers. Investigator planned to compare psychiatric diagnoses, specifically anxiety and depression, with children referred to pediatric clinics.

ELIGIBILITY:
Inclusion Criteria:

* Having psychogenic cough for study group.
* Referred to pediatric clinics.

Exclusion Criteria:

* Chronical psychiatric disorder and pediatric disease history for control group.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who were diagnosed as having psychogenic cough between 2015 and 2018 years. Age and gender matched control who don't have any chronical health problems.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Psychiatric disorders | Baseline
  Total rate of psychiatric disorders, specifically internalizing disorders, identified via semi-structured diagnostic interview

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman Cahid Orengul, Study Director — Bezmialem University Department of Child and Adolescent Psychiatry
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No